CLINICAL TRIAL: NCT00568672
Title: Optimal Duration of Olanzapine Add-on Therapy in Major Depression: a Placebo-controlled, Randomized, Phase III, Pilot Study in Parallel Group Design
Brief Title: Optimal Duration of Olanzapine Add-on Therapy in Major Depression
Acronym: OLA-D
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn because of personal ressources before inclusion of the first patient
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Arnim Quante, Head of Affective Disorders Section, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-000512-82
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Relapse Rate of a Major Depressive Episode; Safety of Olanzapine in Subjects With Major Depression
Keywords: Major Depression; Olanzapine; add-on therapy; antidepressant; atypical antipsychotic
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Olanzapine 5 mg / day
  Interventions: Drug: Olanzapine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5 mg / day for 6 months
  Other Names: EU/1/96/022/002+019

SUMMARY:
Evaluation of olanzapine versus placebo in the continuation therapy of subjects with major depression who had a response with additional olanzapine to an antidepressant.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age 18 - 80
* diagnosis of major depression according dsm-iv, unipolar course
* Hamilton-Depression-Rating-Scale (17 item score) > 18 prior to inclusion
* response towards therapy with antidepressant and olanzapine as defined > 50 % reduction of HAMDD score
* negative pregancy test
* highly effective contraceptive method in women
* no participation in other trial according to German Drug Laq
* normal liver function

Exclusion Criteria:

* pregnancy, lactation
* depressive episode secondary to somatic disease or substance dependency
* contraindication for olanzapine
* treatment with interacting substances (CYP1A2 inhibitors or inductors)
* comorbidity according to DSM-IV, axis I
* denail of consent
* hospital treatment by legal order
* hepatic insufficiency
* severe neurological or medical disease
* adipositas permagna
* HIV-infection
* active viral hapatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10 (Estimated); Primary Completion 2008-01 (Estimated); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Relapse Rate, Hamilton Depression Rating Scale (17 item version) | 6 months

SECONDARY OUTCOMES:
Safety and side effect scales (SWN Scale, CGI), Beck Depression Inventory | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ion Anghelescu, MD, Principal Investigator — Charité - University Berlin, Campus Benjamin Franklin, Department of Psychiatry and Psychotherapy; Arnim Quante, MD, Principal Investigator — Charite, University Berlin, Campus Benjamin Franklin, Department of Psychiatry and Psychotherapy
Locations (1):
- Departement of Psychiatry and Psychotherapy, Charite, University Medicine Berlin, Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- See also: Related Info — https://psychiatrie.charite.de/